CLINICAL TRIAL: NCT04049682
Title: STaRtS: Start Times and Restful Sleep
Brief Title: Start Times and Restful Sleep
Acronym: STaRtS
Status: Withdrawn | Type: Observational
Why Stopped: Study never recruited subjects
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Associate Professor of Medicine, University of California, San Diego
Other Study IDs: 191306
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Excessive Daytime Somnolence; Sleep Deprivation
Keywords: Sleep; Sleep Deprivation; School
MeSH Terms: conditions — Disorders of Excessive Somnolence; Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre Time-change: Daily activity, sleep duration, subjective sleepiness, and response time before change in school start time
- Post Time-change: Daily activity, sleep duration, subjective sleepiness, and response time after change in school start time
  Interventions: Behavioral: Delayed School Start Time

INTERVENTIONS:
Behavioral: Delayed School Start Time — Francis Parker High School implemented 45-minute later school start time.
  Groups: Post Time-change

SUMMARY:
The purpose of this study is to evaluate the efficacy of later school start times in increasing student sleep, and examine the association between later start times and physical activity, screen time, and commute time. Subjects will wear a FitBit activity tracker wristband for two separate 3-month periods (the year before and the year after the Francis Parker High School start time change in the Fall of 2020) and be advised to wear it as much as possible, especially while sleeping or performing physical activity. At the beginning and end of each study period (at 4 occasions), subjects will fill out a few short, non-invasive surveys about their commute, after-school activities, sleepiness, and preferences for morning or evening, and perform the non-invasive psychomotor vigilance test to measure alertness.

DETAILED DESCRIPTION:
Visit 1: Fall 2019, Enrollment and baseline measurements After obtaining informed consent from the parent and assent from the student, baseline data will be obtained. Visit #1 will take place on campus during free periods, lunch or immediately after school and would not interfere with studies. This will include basic demographic data (age, gender) and a questionnaire asking about their average commute time and type, their afterschool activities, as well as an Epworth Sleepiness scale and validated survey of chronotype (Horne-Ostenberg). Subjects will also undergo a standard 10-minute Psychomotor Vigilance Test (PVT) and be given a FitBit. Investigators will assist them in installing the FitBit app and a screen time app, Moment for on their phones. Including the informational part of this visit, enrollment and questionnaires will take about an hour.

Of note, neither the app nor the FitBit will collect geolocalized data. The app does not track and record content, but only gives us the number of minutes per day the phone is on. There is no cost for the app nor does it use cellular data or wireless connection. The data will be collected during study visits rather than in real time.

At this meeting, subjects will be instructed to wear their FitBits as much as possible, especially while sleeping or during physical activity, and to make sure that the screen time app is working on their phone. The investigators recognize that the students will not likely be able to wear their FitBit at all times, but investigators will ask them to use their devices as much as possible. Periodic email communications will be sent out every other week reminding them to continue wearing their FitBit.

Visit 2: Winter 2019, 12-week time point and FitBit collection. Investigators plan to end the study period on December 19, 2019, the Thursday before students go on winter vacation. Depending on when investigators start the study, this would be about 12 weeks after the beginning of the study period (including a non-school week and a few long weekends). At this visit, investigators will repeat all study procedures from visit 1. Investigators will collect the FitBits, facilitate the export of screen time data and allow them to delete the Moment app on their phones. Subjects will be instructed to look for further communications from us at the beginning of the next year. This visit will likely take about 30 minutes.

Visit 3: Fall 2020, Start time change, FitBit redistribution. Francis Parker will switch to a 45 minute later start time for the 2020-21 school year. On the same week of school as the first visit, investigators will hold a meeting in which subjects will repeat all study procedures as in visit 1 Subjects will be given the same FitBit as subjects used in the last study period. Investigators will supervise them as subjects install the FitBit and Moment app on their phones. This visit will likely take about 30 minutes.

At this meeting, subjects will again be instructed to wear their FitBits as much as possible, especially while sleeping or during physical activity, and to make sure that the screen time app is working on their phone. The Periodic email communications will again be sent out every week reminding them to continue wearing their FitBit.

Visit 4: Winter 2020, 12 week time point, final collection. Again, the study period will end on the Thursday before the students go on winter vacation, about 12 weeks from the beginning of the study period. Subjects will fill out another Epworth Sleepiness scale and undergo a PVT, and undergo a brief survey on their perception of how the start time change has affected their sleep and well-being. Investigators will collect FitBits and instruct subjects to delete the Moment app on their phones.

Data Collection and Analysis Epworth and PVT data will be collected and scored according to the standard guidelines for each battery, and our own surveys will be aggregated and analyzed. Moment data is exported as a CSV file which can be opened with Excel.

The information from the FitBit devices will be obtained via Fitabase (a FitBit partner) , which is a data platform designed to aggregate information from FitBits for research purposes. The FitBit device collects and stores information about an individual's activity; this information is automatically synced (e.g., up to every 10-20 minutes when the smartphone's Bluetooth capability is enabled) with the user's smartphone via the FitBit smartphone application using Bluetooth technology. This data is concurrently transmitted to FitBit servers. For subjects enrolled in research studies, Fitabase collects the information from the FitBit servers in near real time and aggregates the information. Investigators can access this data using a secure login provided by Fitabase. A document with more detail on Fitabase security is included with this application.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 or older.
* Enrolled as a freshman, sophomore, or junior at Francis Parker High School.
* In possession of a smartphone compatible with the mobile applications used for the study

Exclusion Criteria:

* Under 13 years old
* Over 19 years old

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 40 High school students (freshmen, sophomores, and juniors during the 2019-20 school year) primarily younger than 18 years old, enrolled at Francis Parker High School
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Daily Activity | 6 months
  Physical activity levels in the form of step counts from FitBit data over two distinct 3-month periods
Sleep Duration | 6 months
  Bedtimes and sleep durations using FitBit data over two distinct 3-month periods

SECONDARY OUTCOMES:
Subjective Sleepiness | 20 minutes
  A subjective measure of daytime sleepiness, measured as an Epworth Sleepiness Score using a questionnaire (Epworth Sleepiness Scale) that combines.
  The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Response Time | 20 minutes
  Reaction times measured in milliseconds using the psychomotor vigilance test.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Owens, MD, Principal Investigator — UCSD
Locations (2):
- United States (2):
  - University of California, San Diego, San Diego, California
  - Francis Parker High School, San Diego, California

IPD SHARING:
Plan to Share IPD: No